CLINICAL TRIAL: NCT06214793
Title: A Phase II Study of Taletrectinib in Previously Treated Metastatic CDH1-mutated Invasive Lobular Cancer (ILC) of the Breast (TaCe)
Brief Title: Taletrectinib in Previously Treated Metastatic CDH1-mutated Invasive Lobular Cancer (ILC)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Anheart acquired by Nuvation Bio; leadership not moving forward
Sponsor: Megan Kruse, MD (Other)
Collaborators: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Megan Kruse, MD, Principal Investigator, MD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5123
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — taletrectinib

STUDY DESIGN:
Intervention Model Description: Single arm, prospective phase II study of taletrectinib in participants with CDH1-mutated breast metastatic ILC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Taletrectinib (Experimental): Taletrectinib 600mg will be given po daily every day within 2 hours of meals on days 1-21, on a 21-day cycle. Study drug will be given until intolerance, consent withdrawal, progression per RECIST 1.1, or death (i.e., no maximum number of cycles).
  Interventions: Drug: Taletrectinib

INTERVENTIONS:
Drug: Taletrectinib — Taletrectinib (AB-106/DS-6051b) is a potent, highly selective, orally bioavailable ROS1 and TRK family inhibitor, which has activity against mutations conferring resistance to crizotinib including in vitro and in vivo against the acquired ROS1 G2032R solvent front mutation. Taletrectinib has been shown to have anti-tumor activity against recombinant ROS1, NTRK1, and NTRK3 in sub-nanomolar concentration in an ATP dependent manner, in addition to completely inhibiting ACK, ALK, DDR1 and LTK at micromolar concentrations. Anti-tumor activity of taletrectinib was observed in two ROS1 rearranged lung cancer cell lines, glioblastoma cell line, and in NTRK-rearranged colorectal cancer cell lines.
  Other Names: AB-106

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of talectrectinib as treatment for Stage IV ILC with CDH1 mutation

DETAILED DESCRIPTION:
Invasive lobular cancer (ILC) represents 10-15% of all breast cancers, up to 75% of ILCs carry a mutation in CDH1 gene which encodes for e-cadherin (ECAD), which is a cell adhesion glycoprotein. Preclinical data using patient derived xenografts have shown loss of ECAD due to CDH1 mutation is associated with an upregulation ROS1 activity, and ROS1 inhibitors have demonstrated synthetic lethality in CDH1-mutated cell lines. Taletrectinib is a novel ROS1/NTRK inhibitor with demonstrated activity in ROS1 mutated non-small cell lung cancer. The purpose of the trial is to estimate the activity of taletrectinib in previously treated CDH1-mutated metastatic breast ILC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. History of histologically or cytologically confirmed diagnosis invasive lobular carcinoma and current diagnosis of metastatic breast cancer
3. Presence of CDH1 mutation as confirmed by any commercially available next generation sequencing (NGS) testing on tumor tissue or liquid biopsy specimens
4. Negative HER2 testing (IHC 1+ or 2+ with negative FISH)
5. Prior Therapy requirements:

   1. For estrogen receptor positive (ER+) participants: prior endocrine therapy with a CDK4/6 inhibitor and at least 1 chemotherapy or antibody drug conjugate in the metastatic setting
   2. For estrogen receptor negative (ER-) participants: at least 2 prior lines of chemotherapy or antibody drug conjugate received in the metastatic setting
6. Participants with central nervous system (CNS) involvement, including leptomeningeal carcinomatosis, which is stable (either asymptomatic or previously treated and controlled are allowed as follows:

   1. Seizure prophylaxis is permitted with non-enzyme-inducing anti-epileptic drugs (non- EIAEDs).
   2. Corticosteroid treatment at a stable or decreasing dose of ≤10 mg prednisone or equivalent if required within 7 days prior to the first dose of taletrectinib.
   3. Local therapy including but not limited to whole brain radiation or gamma knife irradiation treatment must be completed at least 14 days before enrollment and the participant clinically stable (e.g., no corticosteroids or anticonvulsant treatment) for 7 days prior to first dose of taletrectinib (for participants with neurological symptoms or signs due to CNS metastasis at screening).
7. At least 1 measurable lesion per RECIST 1.1 assessed by investigator.
8. Eastern Cooperative Oncology Group Performance Status: 0-2
9. Participant with a life expectancy ≥12 weeks based on the judgement of investigator.
10. Participant with adequate organ function meeting the following criteria:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤3.0 × upper limit of normal (ULN) (or ≤5.0 × ULN, for participants with concurrent liver metastases)
    2. Serum total bilirubin: ≤1.5 × ULN (≤3.0 × ULN for participants with Gilbert syndrome or if liver function abnormalities are due to underlying malignancy)
    3. Absolute neutrophil count: ≥1,000/μL
    4. Platelet count: ≥100,000/μL
    5. Hemoglobin: ≥9.0 g/dL
    6. Estimated creatinine clearance (CrCl) ≥45 mL/min as calculated using the method standard for the institution (eg. Cockcroft - Gault Equation)
11. Males and/or females who meet any of the following criteria:

    1. For males (irrespective of surgical sterilization [vasectomy]): agree to use effective contraception methods during the study intervention period and for at least 90 days after the last dose of investigational drug or agree with complete abstinence.
    2. Females without menses for at least 1 year prior to screening or documented to be surgically sterilized. Women of childbearing potential (WOCBP) must agree to use one highly effective method of contraception or agree with complete abstinence from sexual intercourse since the informed consent until 45 days after the last dose of investigational drug.
12. For all females of childbearing potential, a negative pregnancy test must be obtained within 7 days before starting study treatment. Female participants of non-childbearing potential must meet at least 1 of the following criteria:

    1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state.
    2. Have undergone a documented hysterectomy and/or bilateral oophorectomy.
    3. Have medically confirmed ovarian failure. All other female participants (including female participants with tubal ligations) are considered to be of childbearing potential.
13. The participant is willing and capable to give written informed consent.
14. The participant is willing and capable to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
15. The participant is willing and capable to comply with study site's COVID-19 policies.

Exclusion Criteria:

1. Treatment with small molecule anticancer therapy including other investigational agents or cytotoxic systemic anticancer therapy within 2 weeks (or 5 half-lives of the compound, whichever is shorter) prior to the first dose of taletrectinib; Treatment with immuno-oncology (IO) including immune checkpoint inhibitors within 4 weeks before the first dose of taletrectinib.
2. Major surgical procedure, open biopsy, or significant traumatic injury ≤4 weeks before the first dose of taletrectinib.

   a) Placement of vascular access device is not considered major surgery. Other minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
3. Radiotherapy within 14 days before study treatment. Stereotactic radiosurgery (SRS), stereotactic radiation therapy (SRT), and palliative radiation outside the chest and brain are allowed but must be completed 1 week before starting study treatment.
4. Have been diagnosed with another primary malignancy except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
5. Adverse events due to prior therapy are unresolved to ≤ CTCAE Grade 1 or has not returned to baseline, at the time of the first dose of taletrectinib except for AEs not constituting a safety risk to the patient based on the judgment of investigators.
6. Participants with untreated spinal cord compression caused by tumor and/or cancerous meningitis.
7. History or evidence of interstitial fibrosis, interstitial lung disease or drug-induced pneumonitis (Excluding clinically insignificant or asymptomatic post-radiation pneumonitis).
8. Any gastrointestinal disorders that may affect absorption of oral medications.
9. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV), hepatitis C virus (HCV), or severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.

   Note that the following are permitted:
   1. Participants treated for hepatitis C (HCV) or HIV with no detectable viral load; for at least 1 month prior to the first dose of taletrectinib.

      Note: caution with drug-drug interactions of concomitant anti-HIV agents and CYP3A substrates.
   2. Participants with known hepatitis B (HBV) infections:

   i. with past or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of hepatitis B surface antigen [HBsAg]);

   or

   ii. with inactive HBV carrier state (defined as HBsAg-positive, with normal ALT, and HBV DNA <2,000 IU/mL or <10,000 copies/mL).

   Note: Please consider that for participants in an inactive HBV carrier state or with a resolved HBV infection, there may be a risk of HBV reactivation and anti-HBV prophylaxis should be considered.
10. Clinically significant cardiovascular diseases within 3 months prior to the first dose of talectrectinib: myocardial infarction, severe/unstable angina, coronary/peripheral endovascular treatment, heart failure or cerebrovascular disorder including transient ischemic attack.
11. Ongoing cardiac dysrhythmias of ≥ CTCAE Grade 2, uncontrolled atrial fibrillation of any grade, or QT interval corrected for heart rate by Fredericia's formula (QTcF) >470 milliseconds, or symptomatic bradycardia <45 beats per minute; patient has family or medical history of long QT syndrome.
12. Pregnancy or lactation/breastfeeding.
13. Use of food or drugs that are known potent cytochrome P450 3A4/5 (CYP3A4/5) inhibitors or inducers or P-glycoprotein inhibitors or inducers within 14 days prior to the first dose of study treatment and while on treatment.
14. Administration of agents with potential QT interval prolonging effect within 14 days prior to first dose of study treatment and while on treatment.
15. Participants with other severe medical or mental diseases in whom the risk is increased by the participation to the study or treatment with study treatment in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as measured by RECIST v1 | 24 Weeks
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence.

SECONDARY OUTCOMES:
Progression Free Survival Rate(PFS) | Every 12 weeks until 180 days from EOT until death, withdrawal of informed consent, loss of follow-up or termination of the study by the sponsor, whichever occurs first.
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Clinical Benefit Rate | Up to 6 months (180 days) after completion of therapy or until death, whichever comes first
  Clinical benefit rate as measured by total number of participants with complete response, partial response and stable disease in participants treated with taletrectinib
Duration Of Response(DOR) | Up to 6 months (180 days) after completion of therapy or until death, whichever comes first
  Defined as the subset of participants who achieved a confirmed CR or PR from the date of first documentation of objective response (CR or PR) to the date of first documentation of progressive disease (PD).
Safety analysis, with toxicities graded according to NCI CTCAE v5.0 | Up to 30 days after the final dose of the study drug
  Incidence tables will be generated to summarize incidence of participants reporting at least one episode of each specific adverse event, incidence of adverse events causing withdrawals and incidence of serious adverse events. Listing of adverse events by participants will include the time to onset, the duration of each event, the severity of each event, and the relationship of the event to study therapy, whether it was a serious event, and whether it caused withdrawal. Proportion and exact confidence boundaries (95% CI) will be estimated for toxicity.
Overall Quality Of Life(QOL) with EORTC QLQ-C30 assessments | Assessed every 12 weeks starting from first treatment visit till EOT and then every 12 weeks until 6 months after EOT
  The EORTC QLQ-C30 questionnaire is a 30-item cancer-specific questionnaire that incorporates 5 functioning scales (physical, role, cognition, emotional, and social), 8 symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, loss of appetite, constipation, diarrhea), financial well-being scale and a global scale (based on 2 items: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?").
Overall Quality Of Life(QOL) with FACT-B assessments | Assessed every 12 weeks starting from first treatment visit till EOT and then every 12 weeks until 6 months after EOT
  The FACT-B v4.0 is a 37-item self-reported instrument designed for participants to report on quality of life measures within 5 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Breast Cancer Subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Kruse, Principal Investigator — Cleveland Clinic Foundation, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Marone Cancer Center Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be shared via peer-reviewed publication as a combined summary. Any individual outcomes published per subject will be deidentified utilizing the subject ID (eg. Dose level, demographics, adverse events etc.)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data included in the peer reviewed publication will be publicly available. No raw data will be shared
Access Criteria: A peer-reviewed publication will be made available according to the publishing journal's specifications. CCF personnel will not share study data apart from that which has been published publicly.
URL: http://pubmed.ncbi.nlm.nih.gov/